CLINICAL TRIAL: NCT03802487
Title: A Phase 1, Single-Center, Open-Label, Two-Period, One-Sequence, Single Dose Study to Determine the Absolute Bioavailability of Sotagliflozin in Healthy Male and Female Subjects
Brief Title: Study To Determine Bioavailability of Sotagliflozin in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKM15402; 2017-004937-94 (EudraCT Number); U1111-1200-2077 (Other: UTN)
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus; Healthy Subjects
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Charcoal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sotagliflozin (Experimental): One treatment period includes a single oral dose of sotagliflozin + IV microdose 14C-sotagliflozin tracer plus charcoal. The other treatment period includes a single oral dose of sotagliflozin + IV microdose 14C-sotagliflozin tracer without charcoal.
  Interventions: Drug: Sotagliflozin (SAR439954); Drug: 14C-microtracer; Drug: Charcoal

INTERVENTIONS:
Drug: Sotagliflozin (SAR439954) — Pharmaceutical form: Tablet
  Route of administration: Oral
Drug: 14C-microtracer — Pharmaceutical form: Solution for injection
  Route of administration: Intravenous
Drug: Charcoal — Pharmaceutical form: Granules for suspension
  Route of administration: Oral

SUMMARY:
Primary Objective:

To assess the absolute bioavailability of sotagliflozin via administration of an intravenous (IV) microdose of a 14C-sotagliflozin tracer on top of a single oral dose of unlabeled sotagliflozin without charcoal administration

Secondary Objectives:

* To assess the PK of sotagliflozin and its main metabolite sotagliflozin-3-O-glucuronide (M19) after a single oral dose of sotagliflozin and an IV microdose of a 14C-sotagliflozin tracer without charcoal administration
* To assess the safety and tolerability of single doses of sotagliflozin when administered with and without charcoal

DETAILED DESCRIPTION:
Study duration per participant is up to 54 days including a screening period of up to 28 days, period 1 of 8 days, period 2 of 8 days, a washout period of at least 10 days, and a follow up period of 12-16 days.

The oral drug Sotagliflozin is metabolized by the liver and released in the bile juice into the intestine. Ingestion of charcoal a few hours after the drug administration circumvents the re-uptake of the drug from the intestine back into the blood circulation; instead, Sotagliflozin is eliminated with the feces. By comparison of Sotagliflozin drug administration with and without charcoal, the extent of this so-called enterohepatic circulation can be assessed.

ELIGIBILITY:
Inclusion criteria :

* Male or female subjects, between 18 and 55 years of age, inclusive.
* Body weight between 50.0 and 120.0 kg, inclusive, if male, and between 40.0 and 100.0 kg, inclusive, if female, body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive. BMI between 30.0 and 32.0 is acceptable if investigator judges the subject to have a high muscle mass.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs, ECG and laboratory parameters.

Exclusion criteria:

* Any history or presence of clinically relevant abnormalities at screening which could interfere with the objectives of the study or the safety of the subject's participation.
* Blood donation (400 mL) within 3 months before inclusion.
* History or presence of drug or alcohol abuse.
* Smoking regularly more than 5 cigarettes or equivalent per week, unable to stop smoking during the study.

Excessive consumption of beverages containing xanthine bases.

* If female, pregnancy (defined as positive β-Human Chorionic Gonadotropin blood test), breast-feeding.
* Any medication (including St John's Wort) within 14 days before inclusion with the exception of menopausal hormone replacement therapy; any vaccination within last 28 days; any biologics given within last 4 months.
* Any subject in the exclusion period of a previous study.
* Any subject who cannot be contacted in case of emergency.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies.
* Positive result on urine drug screen.
* Positive alcohol test.
* Participation in a study in which radioisotopes were administered or in which subject was exposed to any radiation other than normal background radiation within the 12 months before the screening visit.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameter: Absolute Bioavailability (F) | Baseline to Day 8 of period 1 (without charcoal)
  Absolute Bioavailability (F) will be a composite endpoint and include Area under plasma concentration (AUC) dose normalized for intravenous (IV) 14C-IMP AUClast dose normalized for oral Investigational Medicinal Product (IMP)

SECONDARY OUTCOMES:
Assessment of PK parameter: Area under the curve (AUC) for oral investigational medicinal product (IMP) | Baseline to Day 8 of each period
  Area under the plasma concentration versus time curve extrapolated to infinity for oral IMP
Assessment of PK parameter: AUC for IMP metabolite | Baseline to Day 8 of each period
  Area under the plasma concentration versus time curve extrapolated to infinity for IMP metabolite
Assessment of PK parameter: AUC for IV 14C-IMP | Baseline to Day 8 of each period
  Area under the plasma concentration versus time curve extrapolated to infinity for IV 14C-IMP
Assessment of PK parameter: AUC for 14C-IMP metabolite | Baseline to Day 8 of each period
  Area under the plasma concentration versus time curve extrapolated to infinity for 14C-IMP metabolite
Assessment of PK parameter: Area under curve versus time (AUClast) for oral IMP | Baseline to Day 8 of each period
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time tlast for oral IMP
Assessment of PK parameter: AUClast for IMP metabolite | Baseline to Day 8 of each period
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time tlast for IMP metabolite
Assessment of PK parameter: AUClast for IV 14C-IMP | Baseline to Day 8 of each period
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time tlast for IV 14C-IMP
Assessment of PK parameter: AUClast for 14C-IMP metabolite | Baseline to Day 8 of each period
  Area under the plasma concentration versus time curve
Assessment of PK parameter: Cmax for oral IMP | Baseline to Day 8 of each period
  Maximum plasma concentration observed for oral IMP
Assessment of PK parameter: Cmax for IMP metabolite | Baseline to Day 8 of each period
  Maximum plasma concentration observed for IMP metabolite
Assessment of PK parameter: Cmax for IV 14C-IMP | Baseline to Day 8 of each period
  Maximum plasma concentration observed for IV 14C-IMP
Assessment of PK parameter: Cmax for 14C-IMP metabolite | Baseline to Day 8 of each period
  Maximum plasma concentration observed for 14C-IMP metabolite
Assessment of PK parameter: tmax for oral IMP | Baseline to Day 8 of each period
  Time to reach Cmax for oral IMP
Assessment of PK parameter: tmax for IMP metabolite | Baseline to Day 8 of each period
  Time to reach Cmax for IMP metabolite
Assessment of PK parameter: tmax for IV 14C-IMP | Baseline to Day 8 of each period
  Time to reach Cmax for IV 14C-IMP
Assessment of PK parameter: tmax for 14C-IMP metabolite | Baseline to Day 8 of each period
  Time to reach Cmax for 14C-IMP metabolite
Assessment of PK parameter: t1/2z for oral IMP | Baseline to Day 8 of each period
  Terminal half-life (t1/2z) associated with the terminal slope for oral IMP
Assessment of PK parameter: t1/2z for IV 14C-IMP | Baseline to Day 8 of each period
  Terminal half-life (t1/2z) associated with the terminal slope for IV 14C-IMP
Assessment of PK parameter: Clearance (CL/F) for oral IMP | Baseline to Day 8 of each period
  Apparent total body clearance for oral IMP
Assessment of PK parameter: Clearance (CL/F) for IV 14C-IMP | Baseline to Day 8 of each period
  Apparent total body clearance for IV 14C-IMP
Assessment of PK parameter: Vz/F for oral IMP | Baseline to Day 8 of each period
  Apparent volume of distribution for oral IMP
Assessment of PK parameter: Vz/F for IV 14C-IMP | Baseline to Day 8 of each period
  Apparent volume of distribution for IV 14C-IMP
Assessment of PK parameter: Vdss/F for oral IMP | Baseline to Day 8 of each period
  Apparent volume of distribution at the steady state for oral IMP
Assessment of PK parameter: Vdss/F for IV 14C-IMP | Baseline to Day 8 of each period
  Apparent volume of distribution at the steady state for IV 14C-IMP
Safety: Adverse events | Baseline to Day 8 of each period
  Number of subjects with adverse events including serious, non-serious, and treatment emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site number 8260001, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org